CLINICAL TRIAL: NCT02127398
Title: Fecal Microbiota Transplantation in Refractory Clostridium Difficile Colitis
Brief Title: Stool Transplants to Treat Refractory Clostridium Difficile Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00053348
Record Dates: First submitted 2014-04-18; First posted 2014-04-30 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Clostridium Difficile Colitis
Keywords: C. difficile colitis; fecal microbiota transplantation
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fecal microbiota transplantation (Experimental): fecal microbiota transplantation
  Interventions: Biological: fecal microbiota

INTERVENTIONS:
Biological: fecal microbiota — fecal microbiota in capsule form

SUMMARY:
It has been shown that restoration of the normal makeup of the bowel bacterial population is the most effective way to treat recurrent colitis due to Clostridium difficile. Restoration of the normal bowel bacterial population is best done by transplanting stool from a healthy donor. The investigators wish to transplant stool from healthy donors to treat recurrent C. difficile colitis by incorporating the stool into capsules that are administered by the oral route.

DETAILED DESCRIPTION:
Recurrent colitis due to Clostridium difficile results from disruption of the normal gut flora, and is very difficult to treat. It is now clear that restoration of the normal gut flora is the most effective way to treat recurrent C. difficile colitis. Restoration of the normal gut flora is best done by transplanting stool from a healthy donor, and this is accepted as a superior therapeutic modality for recurrent C. difficile colitis. This fecal microbiota transplantation can be done with direct instillation of the donor stool into the GI tract via a naso-duodenal tube or colonoscope. Recently, a non-invasive method of stool transplantation has been developed where the donor stool is encapsulated and administered in pill form. The investigators would like to use fecal microbiota transplantation with encapsulated stool as a non-invasive therapy for patients with recurrent C. difficile colitis. To qualify, patients must have a history of, at least, 3 episodes of C difficile colitis within the past year or, at least, 2 episodes of C difficile colitis that resulted in hospitalization. Stool samples will be obtained from healthy volunteers who have been screened for infections that can be transmitted via stool, and the investigators will prepare capsules containing processed stool for administration during a single outpatient clinic visit. Patients will be followed closely after administration of the fecal transplant with serial clinic visits, and the primary endpoint will be prevention of any further episodes of C. difficile colitis in the six month period following transplantation. The investigators will also obtain and store stool samples from patients before and after fecal microbiota transplantation for possible future microbiome analyses. The obvious safety concern is the transmission of an infection from the donor. All donors will be carefully screened for high-risk exposures and will undergo testing of both blood and stool to ensure that they are free of infections due to HIV, acute hepatitis A, acute/chronic hepatitis B, hepatitis C, giardiasis, cryptosporidiosis, and Helicobacter pylori.

ELIGIBILITY:
Inclusion Criteria:

* Study entry is open to adults (>18 years old) who have had three of more episodes of Clostridium difficile colitis within the previous 12 months.

Exclusion Criteria:

* Absolute neutrophil count < 500 cells/mm3
* Active infection at other sites (excluding Clostridium difficile) requiring ongoing antibacterial therapy (antiviral or antifungal therapy is acceptable)
* Current or planned cytotoxic chemotherapy within 14 days of the potential fecal transplantation date
* Life expectancy <180 days
* Diagnosis of inflammatory bowel disease (e.g. Crohn's or ulcerative colitis)
* Inability to swallow capsules
* Indwelling nasogastric, orogastric, gastrostomy, or jejunostomy tube
* History of partial or total gastrectomy
* Short gut syndrome requiring total parenteral nutrition
* Pregnancy
* Documented intestinal parasite infection without documentation of appropriate treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2016-04; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recurrent colitis due to Clostridium difficile | six months
  Patients will be followed 1, 7, 28, and 180 days after the treatment and success will be defined as resolution of C. difficile infection without recurrence within a six-month time period. Patients will be assessed by interview and physical exam. Any patients with suspected persisting/recurring C. difficile colitis will undergo further evaluation with a repeat stool C. difficile toxin assay.

SECONDARY OUTCOMES:
Tolerability of oral fecal microbiota transplantation | six months
  We will monitor for side effects during the administration of the fecal microbiota capsules by close observation within the clinic for one hour. All subjects will return 24 hours after administration for repeat examination and for repeat assessment of tolerability using a questionnaire. Symptoms that will be specifically monitored include the patient's subjective measure of nausea, vomiting, abdominal cramping/pain, belching, diarrhea, constipation, and changes in the quantity or quality of stool.
Safety of oral fecal microbiota transplantation | six months
  The main safety concern is for the transmission of infection from the donor to the recipient. At each follow-up visit (1, 7, 28, and 180 days after treatment) subjects will be assessed for any signs or symptoms of infection by history and physical exam. Some of the specific infections that will be considered will be infectious colitis, infection due to Helicobacter pylori, viral hepatitis, and HIV infection. Patients with signs or symptoms of a suspected infection will undergo appropriate workup with blood and/or stool studies.
rate of repeat therapy for C. difficile colitis within 6 months of fecal microbiota transplantation. | six months
  All subjects will return for evaluation with a comprehensive history and physical exam 180 days after fecal microbiota transplantation, and patients will be asked if they have required any form of therapy for C. difficile colitis in the interim.
Rate of hospitalization | six months
Mortality | six months
  Number of people who die
Rate of adverse events | six months
  number of serious AE's occurring within 6 months of transplant

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Cox, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States